CLINICAL TRIAL: NCT02269579
Title: An Open Label Phase II Pharmacokinetic and Pharmacodynamic Assessment of Treatment With CPX-351 (Cytarabine: Daunorubicin) Liposome for Injection in Acute Leukemias and MDS Patients With Moderate Hepatic Impairment
Brief Title: Pharmacokinetic and Pharmacodynamic Assessment of Treatment With CPX-351 (Cytarabine: Daunorubicin) Liposome for Injection in Acute Leukemias and MDS Patients With Moderate Hepatic Impairment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTR0314-208
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Myelodysplastic Syndrome (MDS)
Keywords: Newly Diagnosed AML; Secondary AML; Relapsed/Refractory AML; Relapsed/Refractory ALL
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Recurrence | interventions — CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPX-351 (Experimental): Study Drug CPX-351 will be given intravenously at 100u/m2 on days 1, 3 and 5 by approximately 90 minute infusion.
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351

SUMMARY:
To assess the impact of moderate hepatic impairment on cytarabine and daunorubicin pharmacokinetics and their metabolites following administration of CPX-351.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily sign an informed consent form
* Age ≥ 18 to ≤ 80 years at the time of signing the informed consent form
* Life expectancy of at least 3 months
* Pathological confirmation by bone marrow documenting the following:

  * Newly Diagnosed De novo AML according to WHO criteria except for Acute Promyelocytic Leukemia or patients with known favorable cytogenetics
  * Newly Diagnosed Secondary AML defined as having a history of an antecedent hematologic disorder (myelodysplastic syndromes [MDS], myeloproliferative disease [MPD]or history of cytotoxic treatment for non-hematologic malignancy)
  * Patients with relapsed/refractory AML regardless of cytogenetic risk
  * Patients with relapsed/refractory ALL
  * Patients with MDS (IPSS score ≥ 1.5)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
* Able to adhere to the study visit schedule and other protocol requirements
* Laboratory values fulfilling the following:

  * Serum creatinine ≤ 2.0mg/dL.
  * Hepatic function with a score of 7-9 points according to the Child-Pugh System
  * Serum alanine aminotransferase or aspartate aminotransferase < 3 times the ULN. Note:If elevated liver enzymes are related to disease; contact medical monitor to discuss.
* Cardiac ejection fraction ≥50% by ECHO or MUGA
* Patients with second malignancies in remission may be eligible if there is clinical evidence of disease stability for a period of greater than 6 months off cytotoxic chemotherapy, documented by imaging, tumor marker studies, etc., at screening. Patients maintained on long-term nonchemotherapy treatment, e.g., hormonal therapy, are eligible.
* All men and women must agree to practice effective contraception during the study period if not otherwise documented to be infertile.

Exclusion Criteria:

* Patients with history of and/or current evidence of myocardial impairment (e.g. cardiomyopathy,ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging)
* Newly diagnosed patients with Acute promyelocytic leukemia [t(15;17)] or favorable cytogenetics, including t(8;21) or inv16
* Clinical evidence of active CNS leukemic involvement
* Chemotherapy or other investigational anticancer therapeutic drugs within 1 week prior to study entry. AEs from prior therapy must have resolved or stabilized so that there is no interference with the assessment of efficacy or safety; in the event of rapidly proliferative disease, however, the use of hydroxyurea is permitted up to 12 hours before study entry. Patients with prior bone marrow or stem cell transplant, considered for inclusion, should be discussed with the medical monitor first.
* Any serious medical condition or psychiatric illness that would prevent the patient from providing informed consent
* Patients with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent)
* Active or uncontrolled infection. Patients with any infection receiving treatment (antibiotic,antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥72 hrs. Patients with fevers believed to be due to leukemia or MDS are eligible provided a thorough infection work-up is negative and the patient is clinically and hemodynamically stable.
* Pregnant or lactating women
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-related metabolic disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Total Drug Plasma PK | Pre-dose and up to Day 21 during first induction only
  The following parameters will be determined:Tmax, Cmax, AUC (0-last), AUC (0-inf), AUC (0-tau), Clast/λz, λz, t1/2, Vss and CL

SECONDARY OUTCOMES:
Serum Copper Levels | Pre-dose and up to Day 21 during the first induction only, prior to every course the patient receives, early termination or end of study and 60 day post end of study.
  The following parameters will be determined:Tmax, Cmax, AUC (0-last), AUC (0-inf), AUC (0-tau), Clast/λz, λz, t1/2, Vss and CL
Urine Sampling | Days 5-10 during the first induction only.
Efficacy and Safety | Efficacy and Safety are measured up until the end of study period, SAEs are measured up to 30 days from the end of study period.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Transparency, Study Director — Jazz Pharmaceuticals
Locations (5):
- United States (5):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Shands Cancer Hospital @ University of Florida, Gainesville, Florida
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - John Theurer Cancer Center @ Hackensack Medical University Medical Center, Hackensack, New Jersey
  - Medical College of Wisconsin, Milwaukee, Wisconsin